CLINICAL TRIAL: NCT04296812
Title: Self-Esteem: A Protective Mechanism for Adolescent Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5190499
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Self Esteem; Suicide and Self-harm
Keywords: occupational Therapy; self-esteem intervention; cognitive behavioral therapy; psychoeducation; suicide
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injeti Self-Love Model (Experimental): Psychoeducational intervention focusing improving self-esteem and increasing self-awareness.
  * The session will start with discussion on healthy relationships, self-esteem.
  * A white board will be used in group format and regular 8.5" by 11" paper during individual session to illustrate the Self-Love model and the characteristics and traits that are effected by "self-love and "lack of self-love".
  * At the end of illustration and discussion there will be handout of the "self-love intervention.
  * The session will end by answering questions and emphasizing the importance of having self-awareness of traits that promote low-self-esteem, and finally, strategies to promote and maintain self-esteem.
  Interventions: Behavioral: Self-Love Model

INTERVENTIONS:
Behavioral: Self-Love Model — The model is a visual illustration shaped as a triangle.
  * The bottom left line is title "Zero Self-Love", moving upward are characteristics identified from "zero self-love" along the line.
  * The bottom right side is titled "Self-Love" moving upward are characteristics identified from having "self-love".
  * At the top of the triangle is a circle with the letter "R" within for relationship.
  * Two small lines project horizontally, from the circle, left and right.
  * At the end of the Left line is a circle with the word "break-up" in the middle, surrounded by terms: drugs, alcohol, self-harming, suicide, and sex" as the consequence of "zero self-love".
  * At the end of right line is a circle with the word "break-up" in the middle surrounded by terms: support system, coping skills, spirituality reflection as the consequences of having self-love.
  The strategies being discussed:
  * Exploring self-esteem strategies.
  * Importance of self-worth in relationships.
  * Importance of self-awareness.

SUMMARY:
This study will explore the effects of the Injeti Self-Love Model intervention on adolescents challenged with low-self-esteem leading to self-harming, suicidal thoughts and suicidal attempts. This study will examine the promotion of self-esteem through the Injeti Self-Love Model as a safety measure against "poor behavioral habits" such as intentional self-harming, substance abuse, suicidal thinking and suicide attempt as means to cope. Study participation will include initial screening, self-assessment, occupational therapy self-esteem intervention of one session, with an individual follow-up, along with an interview, and finishing up with a one-month follow-up interview.

The qualitative research is a methodology for investigating and considering the meaning individuals attribute to a significant human experience. The qualitative approach will be structured around a semi-structured interview initiated at the end of the second follow-up session and after 1-month follow-up.

DETAILED DESCRIPTION:
This study uses a mixed method quasi-experimental pretest and posttest design which incorporates characteristics of both qualitative and quantitative approaches The use of the mixed method design approach is to explore an intervention tool which is administered. The study will be conducted in a locked in-patient psychiatric facility on the adolescent unit. Participants will be engaging in two intervention sessions. The first session will be conducted individually or in a group format. The second session will consist of a follow-up individual session.

Participation in this study involves the following: if the subjects meet the inclusion criteria;

* The research team will gather demographic data from the subjects medical chart which will include the following: gender, age, trauma history, family dynamics such as divorced, single parents, foster family, weight and height, residential and town or city of residence.
* Subject will be asked to complete a self-esteem assessment called the Rosenberg Self-Esteem Scale, this will take about 10 minutes.
* Then the subject will be invited to attend the occupational therapy self-esteem treatment session. The self-esteem intervention is already part of the curriculum at Loma Linda University Behavioral Medicine Center on the adolescent unit. If participants meet inclusion criteria and after signing of consents and PHI, and taking the self-assessment the subjects will be invited to join the self-esteem group session and or individual treatment session if they cannot make it to the group session. The self-esteem treatment is based on a psychoeducation process encouraging discussion and focus on self-awareness of ones own self-esteem. During group processing the therapist will provided the handout of the self-love model.
* Within 2 to 3 days of the self-esteem treatment session there will be an individual follow up session to review the intervention. A self-esteem improvement plan handout will be provided, the subject will complete the self-esteem assessment again and will participate in an interview that will be audio recorded. The interview will take approximately 15 minutes.
* Within 40 days of discharge the subjects will be contacted for a follow-up audio-recorded interview which may be conducted via phone, in-person or videoconference. The subject will also complete the self-esteem assessments again. This may take up to 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The sample will consist of up to 70 male and female adolescents.
* Participants must also be English speaking, and are able to read and write in English.
* Ages 14 to 17 admitted to an in-patient psychiatric facility for:

  * suicidal ideation /attempts,
  * destruction to self or others,
  * homicidal ideation
  * Those that are unable to provide for his or her basic needs for food, clothing, or shelter because of a mental disorder.

Exclusion Criteria:

* Presenting with unmanageable symptoms such as psychosis or mania
* cognitive disabilities that prevent a participant from processing
* Behavioral problems that can disrupt the session and or impair safety during the intervention.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Self-esteem | Changes between baseline and 40 days post initial screening.
  The Rosenberg Self-Esteem Scale is a 10-item self-report measure of global self-esteem. It contains 10 statements connected to global feelings of self-worth or self-acceptance. The items are answered on a four-point scale fluctuating from strongly agree to strongly disagree. A score between 15 and 25 is considered normal, while a score less than 15 indicates potential low self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kugel, OTD, OTR/L, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Behavioral Medicine Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No